CLINICAL TRIAL: NCT06102577
Title: Systemic Adverse Effects After Osteopathic Treatment and the Preventive Effect of Vitamin C: Triple-blind Clinical Trial
Brief Title: Systemic Adverse Effects After Osteopathic Treatment and Vitamin C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Medicina Esportiva i Osteopatia, Spain (Other)
Responsible Party: Principal Investigator, Rafael Merino Solis, Dr. Rafael Merino Solis MD., Centre Medicina Esportiva i Osteopatia, Spain
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OMT and Vit.C
Record Dates: First submitted 2023-10-15; First posted 2023-10-26 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Adverse Effects; Ascorbic Acid; Oxidative Stress
Keywords: Osteopathic Medicine; Manipulation, Osteopathic; Adverse effects; Vitamine C; Ascorbic Acid; Oxidative Stress
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient is randomized at the end of the treatment and the person in charge of collecting the data does not know which group each patient belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1gr. Vitamine C (Experimental): Take 1g. of vitamin C at the end of an osteopathic manual treatment
  Interventions: Dietary Supplement: 1gr. Vitamine C
- 1gr.Placebo (Placebo Comparator): Take 1g. of placebo at the end of an osteopathic manual treatment
  Interventions: Other: 1gr Placebo
- control group (Sham Comparator): control
  Interventions: Other: control group

INTERVENTIONS:
Dietary Supplement: 1gr. Vitamine C — Take 1g. of vitamin C at the end of an osteopathic manual treatment
  Arms: 1gr. Vitamine C
Other: 1gr Placebo — ake 1g. of placebo at the end of an osteopathic manual treatment
  Arms: 1gr.Placebo
Other: control group — control
  Arms: control group

SUMMARY:
The goal of this triple-blind randomized clinical trial is to learn about systemic adverse effects in first visit patients who attend an osteopathic medicine center in Barcelona. The main question it aims to answer are:

• Check if there is a relationship between taking vitamin C and the reduction in the appearance of systemic adverse effects after osteopathic treatment (24-72 hours) First-visit patients, at the end of treatment, are asked to enter the study. If they accept, they are administered 1g. of vitamin C, or 1g. placebo or nothing.

If there is a comparison group: Researchers will compare placebo group, control group and intervention group to see if there is a relationship between taking vitamin C and the appearance of systemic adverse effects].

DETAILED DESCRIPTION:
Introduction Systemic adverse effects (SAE) after osteopathic treatment are rarely reported in the scientific literature. There is a consensus in the scientific literature that these adverse effects occur with a certain frequency, without it being clear what the pathophysiology of such effects is. The relationship between free radicals and central sensitization to pain is increasingly evident. Vitamin C is known as a good electron receptor that is used by the body's antioxidant systems to reduce and also has anti-inflammatory properties. The brain has deficiencies in antioxidant systems and vitamin C has a very important role in the control of oxidative stress.

Objective Check if there is a relationship between taking vitamin C and the reduction in the appearance of systemic adverse effects after osteopathic treatment (24-72 hours).

Design Triple-blind randomized clinical trial, where one group was given 1g of vitamin C, another group was given 1g of placebo and the third group was given nothing. From April 1 to May 30, 2022, patients without food allergies or intolerances were recruited. The patients were randomly assigned to the study groups and neither the patient, nor the therapist, nor the person in charge of collecting the data was aware of which group each patient belonged to. Adverse reactions were classified in relation to pain and fatigue. Data collection was carried out through WhatsApp messages to the patients 72 hours after receiving the treatment.

ELIGIBILITY:
Inclusion Criteria:

* first-visit patients
* of legal age,
* without food allergies or intelorenacies
* the ability to receive and send messages via WhatsApp.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Probability of suffering systemic adverse effects | 3 days
  Odds Ratio

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Merino Solis, MD, Principal Investigator — CMosteoesport
Locations (1):
- Medicina Esportiva i Osteopatia, Mollet del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No